CLINICAL TRIAL: NCT05082207
Title: Effect of Ischemic Preconditioning on Dynamic Thiol-disulfide Balance, Randomized Controlled Trial
Brief Title: Ischemic Preconditioning and Thiol-disulfide Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ischemic preconditioning TDH
Record Dates: First submitted 2021-09-26; First posted 2021-10-18 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Tourniquets
Keywords: thiol/disulfide homeostasis; ischemic preconditioning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischaemic preconditioning (RIPC) (Experimental): The group underwent Remote Ischemic Preconditioning.
  Interventions: Other: Remote Ischemic Preconditioning
- Sham Group (Sham Comparator): Sham control group without remote ischemic preconditioning
  Interventions: Other: sham group

INTERVENTIONS:
Other: Remote Ischemic Preconditioning — Three cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure of systolic blood pressure plus 50 mm Hg.
  Other Names: RIPC group
  Arms: Remote Ischaemic preconditioning (RIPC)
Other: sham group — a deflated cuff placed on the upper arm for 30 min
  Arms: Sham Group

SUMMARY:
Various strategies have been proposed to prevent or mitigate the effects of ischemia-reperfusion injury following the use of tourniquets in orthopedic surgery cases. One of them is applying "remote ischemic preconditioning." This randomized controlled trial is planned to evaluate the effectiveness of remote ischemic preconditioning in preventing tourniquet-induced ischemia-reperfusion injury in total knee arthroscopy with dynamic thiol-disulfide homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients who will undergo total knee arthroplasty surgery under elective conditions

Exclusion Criteria:

* emergency operation,
* Underlying neurological disorder,
* Underlying peripheral vascular disease,
* other types of concurrent surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
thiol/disulfide homeostasis | 24th hour after surgery
  Thiol/disulphide homeostasis will be determined at preoperatively and just before the tourniquet opened and at the 1st, 6th and 24th hours after the tourniquet is opened.

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)